CLINICAL TRIAL: NCT04426513
Title: Type of Magnetic Field and the Effects of Rheumatoid Arthritis Treatment
Brief Title: Magnetotherapy in Rheumatoid Arthritis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jolanta Zwolińska (Other)
Responsible Party: Sponsor-Investigator, Jolanta Zwolińska, PhD, University of Rzeszow
Organization: University of Rzeszow (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Magnetotherapy/ RA
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Rheumatoid Arthritis; Hand Rheumatism
Keywords: Magnetotherapy; Rheumatoid arthritis; Hand function
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Magnetic Field Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Only kinesiotherapy (Active Comparator): Patients have only kinesiotherapy of hand without steroid anti-inflammatory drugs and magnetotherapy.
  Interventions: Other: Kinesiotherapy with magnetotherapy
- Kinesiotherapy with bipolar magnetic field (Experimental): Patients have kinesiotherapy of hand and bipolar magnetic field. All patients without steroid anti-inflammatory drugs.
  Interventions: Other: Kinesiotherapy with magnetotherapy
- Kinesiotherapy with unipolar magnetic field (Experimental): Patients have kinesiotherapy of hand and unipolar magnetic field. All patients without steroid anti-inflammatory drugs.
  Interventions: Other: Kinesiotherapy with magnetotherapy

INTERVENTIONS:
Other: Kinesiotherapy with magnetotherapy — Individual kinesiotherapy. Parameters of magnetic field: 7 mT, f= 0-50 Hz, type of impulse: unipolar or bipolar, rectangular pulse

SUMMARY:
Participants with rheumatoid arthritis with recommendation to physiotherapy.

Created 3 study groups:

1. Only kinesiotherapy
2. Kinesiotherapy with unipolar magnetic field
3. Kinesiotherapy with bipolar magnetic field

Kinesiotherapy with magnetic field give better effects than only kinesiotherapy.

DETAILED DESCRIPTION:
Participants with rheumatoid arthritis with recommendation to physiotherapy. All participants have dysfunction and pain of hand.

Inclusion criteria:

1. II ° and III ° of advancement of radiological changes
2. II ° and III ° of advancement of functional changes
3. Remission, low or moderate RA activity: DAS28
4. Medical order

   1. Magnetotherapy and kinesiotherapy
   2. Kinesiotherapy
   3. Consent to participate in the study
   4. Completion of the research program

Exclusion criteria:

1. Additional physiotherapy treatments for the hands
2. Change in type or dose of pharmacotherapy used
3. Taking steroid anti-inflammatory drugs
4. Malaise and side effects in the subject

Outcome Measures:

1. Duration of morning stiffness
2. The degree of severity of morning stiffness
3. Pain intensity assessment (VAS)
4. Test Box & Blocks
5. Measurement of the palmar surface of the hand
6. Measuring the range of motion in the joints of the hand
7. Measurement of compression force in a cylindrical grip
8. Time to maintain maximum pressure during cylindrical grip
9. Hand volume measurement
10. HAQ-20 test

Intervention:

1. Group 1: Only kinesiotherapy
2. Group 2: Kinesiotherapy with bipolar magnetic field
3. Group 3: Kinesiotherapy with unipolar magnetic field

Assessment:

1. Immediately before start therapy
2. Immediately after therapy (10 treatments in 2 weeks)

ELIGIBILITY:
Inclusion Criteria:

* II ° and III ° of advancement of radiological changes
* II ° and III ° of advancement of functional changes
* Remission, low or moderate RA activity: DAS28
* Medical order
* Magnetotherapy and kinesiotherapy
* Kinesiotherapy
* Consent to participate in the study
* Completion of the research program

Exclusion Criteria:

* Additional physiotherapy treatments for the hands
* Change in type or dose of pharmacotherapy used
* Taking steroid anti-inflammatory drugs
* Malaise and side effects in the subject

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from baseline VAS value immediately after therapy
  Pain severity rating scale. only one value. Minimum value is 0, maximum value is 10. The best is 0, the worst is 10.
Health Assesment Questionaire (HAQ) | Change from baseline HAQ value immediately after therapy
  Subjective assesment of level of disability. Value of each of 8 subsections: minimum value 0, maximum value 3. total score is averaged. The best total score is 0, the worst is 3.

SECONDARY OUTCOMES:
Test Box&Blocks | Change from baseline number of blocks immediately after therapy.
  Objective assessment of level of disability of hand. Number of blocks transfer from box 1 to box 2 during 1 minute.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Hedvig Clinical Provincial Hospital No. 2, ul. Lwowska 60, Rzeszów, Subcarpathian, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richmond SJ. Magnet therapy for the relief of pain and inflammation in rheumatoid arthritis (CAMBRA): a randomised placebo-controlled crossover trial. Trials. 2008 Sep 12;9:53. doi: 10.1186/1745-6215-9-53. PMID 18789135
- [Background] Zwolinska J, Gasior M, Sniezek E, Kwolek A. The use of magnetic fields in treatment of patients with rheumatoid arthritis. Review of the literature. Reumatologia. 2016;54(4):201-206. doi: 10.5114/reum.2016.62475. Epub 2016 Oct 5. PMID 27826175
- [Background] Nasonov VA, Murav'ev IuV, Kuz'mina NN. [Can local therapy of joint syndrome with Dolgit cream be used as an alternative to systemic nonsteroid antiinflammatory drugs in rheumatic diseases?]. Ter Arkh. 1998;70(11):64-6. Russian. PMID 9949465
- [Background] Srikesavan C, Williamson E, Cranston T, Hunter J, Adams J, Lamb SE. An Online Hand Exercise Intervention for Adults With Rheumatoid Arthritis (mySARAH): Design, Development, and Usability Testing. J Med Internet Res. 2018 Jun 27;20(6):e10457. doi: 10.2196/10457. PMID 29950288
- [Background] Erol K, Gok K, Cengiz G, Ozgocmen S. Hand functions in systemic sclerosis and rheumatoid arthritis and influence on clinical variables. Int J Rheum Dis. 2018 Jan;21(1):249-252. doi: 10.1111/1756-185X.13044. Epub 2017 Mar 21. PMID 28322506